CLINICAL TRIAL: NCT07096791
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study Evaluating the Efficacy, Safety, and Pharmacokinetics of KH607 in the Treatment of Adult Female Participants With Postpartum Depressive Disorder
Brief Title: A Phase 2 Study to Evaluate Efficacy and Safety of KH607 Tablets in Woman With Postpartum Depression
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chengdu Kanghong Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KH607-40201
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Postpartum Depressive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KH607 (Experimental): Participants receive KH607, 30 milligrams (mg), oral tablets, once daily for 14 days, as tolerated.
  Interventions: Drug: KH607 tablet
- Placebo (Placebo Comparator): Eligible participants receive matching placebo tablets once daily for 14 days.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: KH607 tablet — oral，once daily for 14 days
  Arms: KH607
Drug: placebo — oral，once daily for 14 days
  Arms: Placebo

SUMMARY:
This is a study evaluating the efficacy, and safety of KH607 in 72 participants diagnosed with Postpartum Depressive Disorder.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, parallel-group, placebo-controlled design. Eligible participants were randomized to KH607 group or placebo group for 14 days.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age: 18 to 45 years old (inclusive), female.
2. Participant had a major depressive episode that began no earlier than the third trimester and no later than the first 4 weeks following delivery, as diagnosed by Structured Clinical Interview for Diagnostic and Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) .
3. Participant was <=12 months postpartum.
4. Participant has a Hamilton Rating Scale for Depression (HAM-D) total score ≥26 at screening and Day 1 (prior to dosing).
5. Participant either must have ceased lactating at screening or, if still lactating or actively breastfeeding at screening, must agree to temporarily cease giving breast milk to her infant(s).
6. Fully understand the procedures and sigh the informed consent.

Key Exclusion Criteria:

1. Participant is currently at significant risk of suicide, or has attempted suicide associated with the current episode of MDD.
2. Participant has a history of treatment-resistant depression, defined as persistent depressive symptoms despite treatment with adequate doses of antidepressants from two different classes for an adequate amount of time.
3. Participant has active psychosis.
4. Participant had used modified electroconvulsive therapy (MECT), transcranial magnetic stimulation (TMS), vagus nerve stimulation (VNS), deep brain stimulation (DBS), light therapy, etc. within 1 month prior to Day 1.
5. Subject has a history of sleep apnea.
6. Participant has a medical history of bipolar disorder, schizophrenia, and/or schizoaffective disorder (such as olanzapine, risperidone, quetiapine, aripiprazole, eptifamol, ziprasidone, caliparazine, sodium valproate, lithium carbonate, etc.) within the current major depressive episode.
7. Participant has a clinically significant abnormal 12-lead ECG at the screening or baseline visits. NOTE: mean QT interval calculated using the Fridericia method (QTcF) of >450 msec in males or >470 msec in females will be the basis for exclusion from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the 17-item Hamilton Rating Scale for Depression (HAM-D17) Total Score at Day 15 | Baseline, Day15
  The HAM-D total score comprised a sum of 17 individual item scores.The total score could range from 0 to 52. Higher scores indicated a greater degree of depression.

SECONDARY OUTCOMES:
Change From Baseline in the 17-item Hamilton Rating Scale for Depression (HAM-D17) Total Score at all other time points | Day3,8,21 and 28
Change From Baseline in the Montgomery and Åsberg Depression Rating Scale (MADRS) Total Score at Day 15 and All Other Time Points | Day 3,8,15,21 and 28
  The MADRS was a ten-item diagnostic questionnaire which psychiatrists used to measure the severity of depressive episodes in participants with mood disorders. It was designed as an adjunct to the HAM-D, to be more sensitive than the Hamilton Scale to the changes brought on by antidepressants and other forms of treatment. Each item yielded a score of 0 to 6. The MADRS total score was calculated as the sum of the 10 individual item scores, which ranged from 0 to 60. Higher MADRS scores indicated more severe depression. A negative change from baseline indicated less severe depression. A positive change from baseline indicated more severe depression. The analysis was performed in participants included in Part A of the study.
Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) Total Score at All Time Points | Day 3,8,15,21 and 28
  The 14-item HAM-A was used to rate the severity of symptoms of anxiety. Each of the 14 items was defined by a series of symptoms, and measured both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Scoring for HAM-A was calculated by assigning scores of 0 (not present) to 4 (very severe), with a total score range of 0 to 56. The HAM-A total score was calculated as the sum of the 14 individual item scores. A negative change from baseline indicated less anxiety. A positive change from baseline indicated more anxiety. The analysis was performed in participants included in Part A of the study.
Change From Baseline in Self-Reported Measures of Depressive Symptoms, as Assessed by the Edinburgh Postnatal Depression Scale (EPDS) Total Score | Day 3,8,15,21 and 28
  The EPDS is a self-rated depressive symptom severity scale specific to the perinatal period which consists of 10 individual items. Each item is rated on a 4-point scale ranging from 0 to 3 points. The EPDS total score is calculated as the sum of the 10 individual item scores, ranging from 0 points to 30 points with a higher score indicating more depression. A negative change indicates improvement.
Percentage of Participants With Clinical Global Impression - Severity (CGI-S) Response | Day 3,8,15,21 and 28
  The CGI-S item employed a 7-point Likert scale to measure the overall severtity in the participant's condition.
Percentage of Participants With Clinical Global Impression - Improvement (CGI-I) Response | Day 3,8,15,21 and 28
  The CGI-I item employed a 7-point Likert scale to measure the overall improvement in the participant's condition post-treatment. The investigator rated the participant's total improvement whether or not it was due entirely to drug treatment. The CGI-I was only rated at post-treatment assessments. By definition, all CGI-I assessments were evaluated against baseline conditions. CGI-I response was defined as having a CGI-I global improvement score of 1 (very much improved) or 2 (much improved). The analysis was performed in participants included in Part A of the study. Data is reported for participants who had CGI-I response.
Percentage of Participants With HAM-D Response | Day 3,8,15,21 and 28
  HAM-D response was defined as having a 50% or greater reduction from baseline in HAM-D total score. The analysis was performed in participants included in Part A of the study. Data is reported for participants who had HAM-D response.
Percentage of Participants With HAM-D Remission | Day 3,8,15,21 and 28
  HAM-D remission was defined as having a HAM-D total score of ≤7. The analysis was performed in participants included in Part A of the study.

IPD SHARING:
Plan to Share IPD: Yes